CLINICAL TRIAL: NCT02890030
Title: Sequelae of Treatment in Survivors of Testicular Cancer Creation of a Non-exposed Comparison Group for the Platinum Study
Brief Title: The Platinum Study Comparison Group
Status: Completed | Type: Observational
Sponsor: Lawrence Einhorn (Other)
Responsible Party: Sponsor-Investigator, Lawrence Einhorn, Distinguished Professor of Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Other Study IDs: IRB No. 1604502652
Record Dates: First submitted 2016-06-08; First posted 2016-09-07 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Testicular Neoplasms
Keywords: Cisplatin-based therapy; Ototoxicity; Neurotoxicity
MeSH Terms: conditions — Testicular Neoplasms; Ototoxicity; Neurotoxicity Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Case-Control: Patients with testicular germ cell tumor who were treated with surgery and not cisplatin-based chemotherapy
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — * Neurotoxicity
  * Medications of interest
  * General health
  * Family history

SUMMARY:
The patients enrolled on this new study will serve as an appropriate comparison group consisting of patients with the diagnosis of germ cell testicular cancer who were cured with surgical resection and did not receive cisplatin-based chemotherapy with a group of patients from another study who did receive cisplatin-based chemotherapy.

DETAILED DESCRIPTION:
Primary Objective

To compare the prevalence of ototoxicity and neurotoxicity in GCT cancer survivors who only had surgery to a similar population from The Platinum Study (RSRB45410/1305011509) who received cisplatin-based combination chemotherapy.

Secondary Objective

To compare the prevalence of obesity, hypertension, and use of antidepressants/anxiolytics in GCT cancer survivors who only had surgery to a similar population from The Platinum Study who received cisplatin-based combination chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or confirmation of diagnosis of a histologically or serologically confirmed testicular germ cell tumor (GCT) or GCT at another anatomic location
* Age at GCT diagnosis: 55 years of age or younger
* Males, 18 years of age or older at time of study consent
* Subject is able to provide consent
* Subject is able to speak and read English
* Treatment consisted of surgery only (i.e., orchiectomy and/or retroperitoneal lymph node dissection [RPLND]) for either initial testicular germ cell tumor (GCT) or subsequent testicular cancer
* Subject completed surgery > 1 year ago
* Subject is currently undergoing active follow-up at IU
* Subject did not require any subsequent chemotherapy, salvage chemotherapy treatment or bone marrow transplant.
* Subject had no prior chemotherapy of any kind

Exclusion Criteria:

* Patients with prior chemotherapy (whether for GCT or any other cancer)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male patients with testicular germ cell tumor diagnosis at the age of 18-55 who were treated with surgery only and not chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with ototoxicity | 1 year after surgery
  The proportion of patients from this study will be compared to the proportion of patients with The Platinum Study.
Proportion of patients with neurotoxicity | 1 year after surgery
  The proportion of patients from this study will be compared to the proportion of patients with The Platinum Study.

SECONDARY OUTCOMES:
Proportion of patients with obesity | 1 year after surgery
  The proportion of patients from this study will be compared to the proportion of patients with The Platinum Study.
Proportion of patients with hypertension | 1 year after surgery
  The proportion of patients from this study will be compared to the proportion of patients with The Platinum Study.
Proportion of patients who use antidepressants/anxiolytics | 1 year after surgery
  The proportion of patients from this study will be compared to the proportion of patients with The Platinum Study.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States